CLINICAL TRIAL: NCT04907578
Title: Thromboelastography (TEG) In the Intrauterine Growth Restriction (IUGR) Neonatal Population by Gestational Age
Status: Withdrawn | Type: Observational
Why Stopped: Study will not commence
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jonathan H. Waters, Professor, University of Pittsburgh
Other Study IDs: STUDY21040124
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Intrauterine Growth Restriction
Keywords: Thromboelastography; Intrauterine Growth Restriction; Neonate; Gestational age; hemostasis; coagulopathy
MeSH Terms: conditions — Fetal Growth Retardation; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators plan to collect discarded blood specimens (1-2 mL of placental umbilical vein blood following umbilical cord clamping) in order to perform TEG analysis, in duplicate when possible, immediately following the live birth of a viable neonate. No additional specimens will be collected for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postpartum full term neonates: immediate postpartum full term neonates with no intrauterine growth restricted
- intrauterine growth restricted neonates: preterm or full-term intrauterine growth restricted neonates

SUMMARY:
The investigators aim to improve the understanding of TEG in this population in an effort to improve outcomes in a population at high risk in both the presence and absence of blood product transfusions.

DETAILED DESCRIPTION:
The investigators plan to 1.) examine dynamic hemostasis as measured by TEG in the intrauterine growth restriction (IUGR) neonatal population due to a high risk of requiring blood transfusions, 2.) determine the influence of gestational age on TEG in this population, and 3.) examine the utility of TEG as a tool for identifying coagulopathy in IUGR neonates.

The investigators hypothesize that thromboelastography parameters will change with gestational age in the IUGR population in a manner similar to non-IUGR populations and that neonatal comorbidities, maternal factors, and socioeconomic status will influence TEG values; TEG is likely a useful marker of dynamic hemostasis in this neonatal subpopulation.

ELIGIBILITY:
Inclusion Criteria:

Participants included for medical record data and blood sample collection will be:

* Neonates diagnosed with intrauterine growth restriction, defined as a weight below the estimated 10th percentile and accordingly identified as such in any peripartum evaluation AND
* May have additional comorbidities AND
* Full term IUGR neonates will be have a gestational age of 37 weeks or greater OR
* Preterm IUGR neonates will have a gestational age less than 37 weeks OR
* Preterm IUGR neonates will have a gestational age less than 37 weeks

Participants included for medical record review data collection ONLY will be:

Mothers of eligible neonates

Exclusion Criteria:

* Constitutionally (familial) low birth weight, i.e. small for gestational age, babies OR
* Born to women with life threatening coexisting morbidities (this may include severe pre-eclampsia, diabetes or suspected infections including HIV or herpes) OR
* Neonates with an abnormal delivery or perinatal course including:

Fetal demise, death in the first week after birth, neonatal encephalopathy, meconium aspiration, and physical birth injuries (fractures and brachial plexus injuries)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from Magee-Womens Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Dynamic hemostasis measured by Thromboelastography (TEG) in intrauterine growth restriction (IUGR) neonatal population verse non-IUGR populations | Immediately postpartum
  Discarded blood specimens (1-2 mL of placental umbilical vein blood following umbilical cord clamping) will be needed to perform TEG analysis, in duplicate when possible, immediately following the live birth of a viable neonate. The output of the TEG will include maximum amplitude (mm), which is a reflection of clot strength and a function of the maximum dynamic properties of fibrin and platelet bonding and correlates to platelet function.

SECONDARY OUTCOMES:
Clot formation measured by Thromboelastography (TEG) in intrauterine growth restriction (IUGR) neonatal population verse non-IUGR populations | Immediately postpartum
  Discarded blood specimens (1-2 mL of placental umbilical vein blood following umbilical cord clamping) will be needed to perform TEG analysis, in duplicate when possible, immediately following the live birth of a viable neonate. The output of the TEG will include R time (min), which represents a period of latency from start to initial fibrin formation.
Rate of clot formation measured by Thromboelastography (TEG) in intrauterine growth restriction (IUGR) neonatal population verse non-IUGR populations | Immediately postpartum
  Discarded blood specimens (1-2 mL of placental umbilical vein blood following umbilical cord clamping) will be needed to perform TEG analysis, in duplicate when possible, immediately following the live birth of a viable neonate. The output of the TEG will include α-Angle (degree), which measures the speed at which fibrin build-up and cross-linking takes place, assesses the rate of clot formation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan H. Waters, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Waters JH. The role of viscoelastic testing in the management of the parturient. Transfusion. 2020 Oct;60 Suppl 6:S70-S74. doi: 10.1111/trf.15928. Epub 2020 Jun 22. PMID 32567712
- [Result] Sayce AC, Neal MD, Leeper CM. Viscoelastic monitoring in trauma resuscitation. Transfusion. 2020 Oct;60 Suppl 6:S33-S51. doi: 10.1111/trf.16074. PMID 33089933